CLINICAL TRIAL: NCT06095245
Title: The Outcome of Subthalamic Deep Brain Stimulation in Advanced Parkinson's Disease and Morphometric Differences
Brief Title: The Outcome of Subthalamic Deep Brain Stimulation in Advanced Parkinson's Disease and Morphometry
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Principal Investigator, Maija Koivu, M.D., Specialist in Neurology, Hospital District of Helsinki and Uusimaa
Other Study IDs: 7435
Record Dates: First submitted 2023-09-26; First posted 2023-10-23 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 35 patients with advanced PD treated with subthalamic deep brain stimulation: 35 patients with advanced PD treated with subthalamic deep brain stimulation. The decision of DBS treatment had been performed on the clinical decision by the treating neurologist and the patients. Patients are between 18 and 80 years old.

SUMMARY:
The research will evaluate possible clinical and individual brain topographic features affecting the outcome in subthalamic deep brain stimulation (DBS) with patients with Parkinson's disease (PD). The patient cohort consists 35 PD patients treated with subthalamic DBS in 2020-2022. The clinical features (such as age, disease duration, response to levodopa in the levodopa challenge test) will be evaluated retrospectively from the medical records and brain topographic features from the preoperative 3 Tesla brain imaging.

DETAILED DESCRIPTION:
Subthalamic deep brain stimulation (STN-DBS) is known to enhance motor function in advanced Parkinson's disease and to enable a significant reduction of the use of anti-Parkinsonian medication. A levodopa challenge test is considered as a good predictor of DBS outcome, as well as disease duration. There are heterogenous findings on the age effect on DBS outcome. In recent years, the effect of STN's connectivity with other brain areas on DBS outcome have drawn more attention. The study aim was to evaluate, alongside the clinical predictors, the effect of the patients' individual brain topography on DBS outcome.

The medical records of 35 patients with PD was used to analyze DBS outcome measured with the following scales: Unified Parkinson's Disease Questionnaire, use of anti-Parkinsonian medication (LEDD), Abnormal Involuntary Movement Scale, Beck Depression Inventory, Parkinson's Disease Questionnaire 39, Non-Motor Symptoms Questionnaire. The 3 Tesla preoperative brain MRI images were analyzed with MATLAB for morphometric differences.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Parkinson's disease and subthalamic deep brain stimulation treatment. The DBS screening and operation done in Helsinki University Hospital (HUS)

Exclusion Criteria:

* Patients with Parkinson's disease and not treated with subthalamic DBS in HUS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consists of patients with Parkinson's disease and treated with subthalamic DBS in HUS
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The clinical outcome of subthalamic DBS as evaluated with UPDRS III and levodopa equivalent daily dosage changes | 6 months
  The UPDRS III scores and levodopa equivalent daily dosage at baseline and at 6-month's visit will be evaluated and the changes will be analyzed as clinical outcome of DBS treatment

SECONDARY OUTCOMES:
The patients' individual brain tomographic features affecting the DBS outcome | 6 months
  Whole brain topography and grey matter clusters will be measured using mathlab program and the volumes will be compared to the UPDRS III and LEDD changes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology and department of Neurosurgery Helsinki University Hospital, Helsinki, Finland